CLINICAL TRIAL: NCT03338816
Title: ENVISION: A Phase 3 Randomized, Double-blind, Placebo-Controlled Multicenter Study With an Open-label Extension to Evaluate the Efficacy and Safety of Givosiran in Patients With Acute Hepatic Porphyrias
Brief Title: ENVISION: A Study to Evaluate the Efficacy and Safety of Givosiran (ALN-AS1) in Patients With Acute Hepatic Porphyrias (AHP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-AS1-003
Expanded Access: NCT04056481 (Approved for marketing)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2022-05

CONDITIONS: Acute Hepatic Porphyria; Acute Intermittent Porphyria; Porphyria, Acute Intermittent; Acute Porphyria; Hereditary Coproporphyria (HCP); Variegate Porphyria (VP); ALA Dehydratase Deficient Porphyria (ADP)
Keywords: Acute Intermittent Porphyria (AIP); Acute Hepatic Porphyria (AHP); Hereditary Coproporphyria (HCP); Variegate Porphyria (VP); ALA dehydratase deficient porphyria (ADP) (ALAD); RNAi therapeutic; Porphyria
MeSH Terms: conditions — Coproporphyria, Hereditary; Porphyria, Acute Intermittent; Porphyria, Variegate; Porphyrias | interventions — givosiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Givosiran/Givosiran (Experimental): Givosiran 2.5 mg/kg administered subcutaneously (SC), monthly (QM), for 6 months during the 6-Month Double-blind (DB) Period, followed by givosiran 2.5 mg/kg or 1.25 mg/kg SC, QM for 29 months during the Open-label Extension (OLE) Period.
  Interventions: Drug: Givosiran; Drug: Placebo
- Placebo/Givosiran (Placebo Comparator): Matching placebo (normal saline [0.9% NaCl]) was administered SC, QM, for 6 months during the 6-Month DB Period, followed by givosiran 2.5 mg/kg or 1.25 mg/kg SC, QM for 29 months during the OLE period.
  Interventions: Drug: Givosiran; Drug: Placebo

INTERVENTIONS:
Drug: Givosiran — Givosiran by SC
  Other Names: ALN-AS1; GIVLAARI
Drug: Placebo — Matching placebo (normal saline [0.9% NaCl]) by SC

SUMMARY:
The purpose of this study is to evaluate the effect of subcutaneous givosiran (ALN-AS1), compared to placebo, on the rate of porphyria attacks in patients with Acute Hepatic Porphyrias (AHP).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 12 years of age
* Diagnosed with Acute Hepatic Porphyria (Acute Intermittent Porphyria, Hereditary Corproporhyria, Variegate Porphyria, aminolevulinic acid (ALA) dehydratase deficient porphyria)
* Elevated urinary or plasma porphobilinogen (PBG) or ALA values within the past year,
* Have active disease, with at least 2 documented porphyria attacks within the last 6 months
* Willing to discontinue or not initiate the use of prophylactic hemin throughout the study.
* Women of child bearing potential must have a negative serum pregnancy test, not be nursing, and use acceptable contraception

Exclusion Criteria:

* Clinically significant abnormal laboratory results
* Anticipated liver transplantation
* History of multiple drug allergies or intolerance to subcutaneous injections
* Active HIV, hepatitis C virus, or hepatitis B virus infection(s)
* History of recurrent pancreatitis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (36):
- United States (10):
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Galveston, Texas
  - Clinical Trial Site, Salt Lake City, Utah
  - Clinical Trial Site, Seattle, Washington
- Australia (3):
  - Clinical Trial Site, Parkville, Victoria
  - Clinical Trial Site, Auchenflower
  - Clinical Trial Site, Camperdown
- Clinical Trial Site, Sofia, Bulgaria
- Clinical Trial Site, Edmonton, Canada
- Clinical Trial Site, Odense, Denmark
- Clinical Trial Site, Helsinki, Finland
- Clinical Trial Site, Paris, France
- Germany (2):
  - Clinical Trial Site, Chemnitz
  - Clinical Trial Site, Munich
- Clinical Trial Site, Modena, Italy
- Japan (3):
  - Clinical Trial Site, Hamamatsu
  - Clinical Trial Site, Iizuka
  - Clinical Trial Site, Tokyo
- Clinical Trial Site, Mexico City, Mexico
- Clinical Trial Site, Rotterdam, Netherlands
- Clinical Trial Site, Warsaw, Poland
- Clinical Trial Site, Seoul, South Korea
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, El Palmar
  - Clinical Trial Site, Pamplona
- Clinical Trial Site, Stockholm, Sweden
- Taiwan (3):
  - Clinical Trial Site, Taichung
  - Clinical Trial Site, Taipei
  - Clinical Trial Site, Taoyuan
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232
- [Derived] Lee MJ, Kuo HC, Chou LN, Sweetser MT, Wang JD. A randomized, placebo-controlled study of givosiran in patients with acute hepatic porphyrias (ENVISION): Final (36-month) analysis of the Taiwan Cohort. J Formos Med Assoc. 2024 Jun;123(6):679-686. doi: 10.1016/j.jfma.2023.10.016. Epub 2023 Dec 2. PMID 38044204
- [Derived] Kuter DJ, Bonkovsky HL, Monroy S, Ross G, Guillen-Navarro E, Cappellini MD, Minder AE, Hother-Nielsen O, Ventura P, Jia G, Sweetser MT, Thapar M; ENVISION Investigators. Efficacy and safety of givosiran for acute hepatic porphyria: Final results of the randomized phase III ENVISION trial. J Hepatol. 2023 Nov;79(5):1150-1158. doi: 10.1016/j.jhep.2023.06.013. Epub 2023 Jul 20. PMID 37479139
- [Derived] Wang B, Ventura P, Takase KI, Thapar M, Cassiman D, Kubisch I, Liu S, Sweetser MT, Balwani M. Disease burden in patients with acute hepatic porphyria: experience from the phase 3 ENVISION study. Orphanet J Rare Dis. 2022 Aug 26;17(1):327. doi: 10.1186/s13023-022-02463-x. PMID 36028858
- [Derived] Balwani M, Sardh E, Ventura P, Peiro PA, Rees DC, Stolzel U, Bissell DM, Bonkovsky HL, Windyga J, Anderson KE, Parker C, Silver SM, Keel SB, Wang JD, Stein PE, Harper P, Vassiliou D, Wang B, Phillips J, Ivanova A, Langendonk JG, Kauppinen R, Minder E, Horie Y, Penz C, Chen J, Liu S, Ko JJ, Sweetser MT, Garg P, Vaishnaw A, Kim JB, Simon AR, Gouya L; ENVISION Investigators. Phase 3 Trial of RNAi Therapeutic Givosiran for Acute Intermittent Porphyria. N Engl J Med. 2020 Jun 11;382(24):2289-2301. doi: 10.1056/NEJMoa1913147. PMID 32521132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with acute hepatic porphyrias (AHP) were enrolled at thirty-six sites in Australia, Bulgaria, Canada, Germany, Denmark, Spain, Finland, France, United Kingdom, Italy, Japan, Korea (the Republic of), Mexico, Netherlands, Poland, Sweden, Taiwan and the United States.
Groups:
- Placebo 6-Month DB: Matching placebo (normal saline [0.9% NaCl]) was administered subcutaneously (SC), monthly (QM), for 6 months during the 6-Month Double-blind (DB) Period.
- Givosiran 2.5 mg/kg 6-Month DB: Givosiran 2.5 mg/kg administered SC, QM, for 6 months during the 6-Month DB Period.
- Placebo/Givosiran: Patients who received placebo during the 6-Month DB Period then entered the Open-Label Extension (OLE) Period and were administered givosiran 2.5 mg/kg or 1.25 mg/kg SC, QM for 29 months. Upon implementation of protocol Amendment 5, active patients receiving 1.25 mg/kg givosiran once monthly in the OLE had their dose increased to 2.5 mg/kg givosiran once monthly.
- Givosiran/Givosiran: Patients who received givosiran during the 6-Month DB Period then entered the OLE Period and were administered givosiran 2.5 mg/kg or 1.25 mg/kg SC, QM mg/kg for 29 months. Upon implementation of protocol Amendment 5, active patients receiving 1.25 mg/kg givosiran once monthly in the OLE had their dose increased to 2.5 mg/kg givosiran once monthly.
Period: 6-Month Double-blind Period
Arm/Group | Placebo 6-Month DB | Givosiran 2.5 mg/kg 6-Month DB | Placebo/Givosiran | Givosiran/Givosiran
Started | 46 | 48 | 0 | 0
Completed | 46 | 48 (1 participant discontinued treatment during the 6-month DB period due to an adverse event but completed the 6-month DB Visit) | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 6-Month DB + Open-Label Extension Period
Arm/Group | Placebo 6-Month DB | Givosiran 2.5 mg/kg 6-Month DB | Placebo/Givosiran | Givosiran/Givosiran
Started | 0 | 0 | 46 | 47
Completed | 0 | 0 | 38 | 41
Not Completed | 0 | 0 | 8 | 6
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3
Not completed — Patient Desired Lower Dose | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) consisted of all participants who received at least one dose of study drug.
Groups:
- Placebo: Matching placebo (normal saline [0.9% NaCl]) was administered SC, QM, for 6 months during the 6-Month DB Period, followed by givosiran 2.5 mg/kg or 1.25 mg/kg SC, QM for 29 months during the OLE period.
- Givosiran: Givosiran 2.5 mg/kg administered SC, QM, for 6 months during the 6-Month DB Period, followed by givosiran 2.5 mg/kg or 1.25 mg/kg SC, QM for 29 months during the OLE Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Givosiran | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (10.5) | 40.1 (12.1) | 38.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 34 | 39 | 73
  More than One Race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Porphyria Attacks in Participants With Acute Intermittent Porphyria (AIP)
Description: Porphyria attacks were defined as meeting all of the following criteria: an acute episode of neurovisceral pain in the abdomen, back, chest, extremities and/or limbs, no other medically determined cause, and required treatment with intravenous (IV) dextrose or hemin, carbohydrates, or analgesics, or other medications such as antiemetics at a dose or frequency beyond the participant's usual daily porphyria management. The annualized rate of porphyria attacks is a composite endpoint which included porphyria attacks requiring hospitalization, urgent healthcare visit, or IV hemin administration at home.
Time Frame: 6 months
Population: AIP participants in the Full Analysis Set (FASAIP): All randomized AIP participants (with identified mutation in the hydroxymethylbilane synthase [HMBS] gene) who received at least one dose of study drug.
Measure: Mean (95% Confidence Interval); unit: annualized attack rate
Groups:
- Placebo: Matching placebo (normal saline [0.9% NaCl]) was administered SC, QM, for 6 months during the 6-Month DB Period.
- Givosiran 2.5 mg/kg: Givosiran 2.5 mg/kg administered SC, QM, for 6 months during the 6-Month DB Period.
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
annualized attack rate | 12.52 [9.35 to 16.76] | 3.22 [2.25 to 4.59]
Statistical Analysis 1: Comparison: Placebo vs Givosiran 2.5 mg/kg; Negative binomial regression model with treatment group and stratification factors (prior hemin prophylaxis status and historical attack rates) as fixed effects and the logarithm of the follow-up time as an offset variable; Test type: Superiority; p < 0.0001, Negative binomial regression model — P=6.040E-09; Rate ratio = 0.26, 95% CI 2-sided [0.16 to 0.41]

2. Secondary Outcome: The Pharmacodynamic (PD) Effect of Givosiran on Urine Levels of Delta-aminolevulinic Acid (ALA) in Participants With AIP
Description: The PD effect of givosiran was evaluated by spot urine ALA levels normalized to spot urine creatinine levels.
Time Frame: 3 and 6 months
Population: FASAIP: All randomized AIP participants (with identified mutation in the HMBS gene) who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmol/mol creatinine (Cr)
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
mmol/mol creatinine (Cr)
  Month 3 | 19.965 (1.475) | 1.756 (1.413)
  Month 6 | 23.150 (2.534) | 4.013 (2.352)

3. Secondary Outcome: The PD Effect of Givosiran on Urine Levels of Porphobilinogen (PBG) in Participants With AIP
Description: The PD effect of givosiran was evaluated by spot urine PBG levels normalized to spot urine creatinine levels.
Time Frame: 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/mol Cr
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
mmol/mol Cr | 49.110 (4.959) | 12.906 (4.642)

4. Secondary Outcome: Annualized Rate of Hemin Administration in Participants With AIP
Description: Annualized rate of hemin doses was evaluated as annualized days of hemin use.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: annualized rate of use
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
annualized rate of use | 29.71 [18.41 to 47.94] | 6.77 [4.20 to 10.92]

5. Secondary Outcome: Annualized Rate of Porphyria Attacks in Participants With AHP
Description: as for outcome 1
Time Frame: 6 months
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of study drug.
Measure: Mean (95% Confidence Interval); unit: annualized attack rate
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 46 | 48
annualized attack rate | 12.26 [9.22 to 16.29] | 3.35 [2.37 to 4.74]

6. Secondary Outcome: Area Under the Curve (AUC) of the Change From Baseline in Weekly Mean Score of Daily Worst Pain as Measured by the Brief Pain Inventory-Short Form (BPI-SF) Numeric Rating Scale (NRS) in Participants With AIP
Description: Participants rated worst daily pain score in an eDiary using the 11-point BPI-SF NRS, in which 0=no pain and 10=worst pain. Daily eDiary entries were averaged into a weekly (i.e. 7 day) score. The change from baseline in weekly mean scores is defined as the post baseline weekly mean score minus the baseline score. Lower scores indicate an improvement. The 6-month AUC was calculated based on change from baseline in weekly mean scores.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale*week
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale*week | 5.286 [-23.048 to 11.145] | -11.514 [-29.181 to 3.040]

7. Secondary Outcome: Average Change From Baseline in Weekly Mean Score of Daily Worst Pain as Measured by the Brief Pain Inventory-Short Form (BPI-SF) Numeric Rating Scale (NRS) in Participants With AIP
Description: Participants rated worst daily pain score in an eDiary using the 11-point BPI-SF NRS, in which 0=no pain and 10=worst pain. Daily eDiary entries were averaged into a weekly (i.e. 7 day) score. The change from baseline in weekly mean scores is defined as the postbaseline weekly mean score minus the baseline score. Lower scores indicate an improvement.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale | 0.245 [-1.020 to 0.470] | -0.506 [-1.309 to 0.143]

8. Secondary Outcome: AUC of the Change From Baseline in Weekly Mean Score of Daily Worst Fatigue Score as Measured by the Brief Fatigue Inventory-Short Form (BFI-SF) NRS in Participants With AIP
Description: Participants rated daily worst fatigue score in an eDiary using the 11-point BFI-SF NRS, in which 0=no fatigue and 10=worst fatigue. Daily eDiary entries were averaged into a weekly (i.e. 7 day) score. The change from baseline in weekly mean scores is defined as the post baseline weekly mean score minus the baseline score. Lower scores indicate an improvement. The 6-month AUC was calculated based on change from baseline in weekly mean scores.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale*week
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale*week | -4.208 (4.689) | -11.148 (4.501)

9. Secondary Outcome: Average Change From Baseline in Weekly Mean Score of Daily Worst Fatigue Score as Measured by the Brief Fatigue Inventory-Short Form (BFI-SF) NRS in Participants With AIP
Description: Participants rated daily worst fatigue score in an eDiary using the 11-point BFI-SF NRS, in which 0=no fatigue and 10=worst fatigue. Daily eDiary entries were averaged into a weekly (i.e. 7 day) score. The change from baseline in weekly mean scores is defined as the postbaseline weekly mean score minus the baseline score. Lower scores indicate an improvement.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale | -0.182 (0.209) | -0.502 (0.200)

10. Secondary Outcome: AUC of the Change From Baseline in Weekly Mean Score Daily Worst Nausea Score as Measured by NRS in Participants With AIP
Description: Participants rated worst daily nausea score in an eDiary using an 11-point NRS, in which 0=no nausea and 10=worst nausea. Daily eDiary entries were averaged into a weekly (i.e. 7 day) score. The change from baseline in weekly mean scores is defined as the postbaseline weekly mean score minus the baseline score. Lower scores indicate an improvement. The 6-month AUC was calculated based on change from baseline in weekly mean scores.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale | -4.011 (3.453) | 1.481 (3.310)

11. Secondary Outcome: Average Change From Baseline in Weekly Mean Score Daily Worst Nausea Score as Measured by NRS in Participants With AIP
Description: Participants rated worst daily nausea score in an eDiary using an 11-point NRS, in which 0=no nausea and 10=worst nausea. Daily eDiary entries were averaged into a weekly (i.e. 7 day) score. The change from baseline in weekly mean scores is defined as the postbaseline weekly mean score minus the baseline score. Lower scores indicate an improvement.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale | -0.181 (0.154) | 0.067 (0.147)

12. Secondary Outcome: Change From Baseline in the Physical Component Summary (PCS) of the 12-Item Short Form Survey (SF-12) in Participants With AIP
Description: The SF-12 is a survey designed for use in patients with multiple chronic conditions. This 12-item scale can be used to assess the physical and mental health of respondents. 10 of the 12 questions are answered on a 5 point likert scale and 2 are answered on a 3 point likert scale. The questions are then scored and weighted into 2 subscales, physical health and mental health. Respondents can have a score that ranges from 0-100 with 100 being the best score and indicating high physical or mental health. A 3 point change in SF-12 score reflects a meaningful difference. A higher score indicates improvement.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Givosiran 2.5 mg/kg
Number analyzed (Participants) | 43 | 46
score on a scale | 1.431 (1.220) | 5.369 (1.169)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through completion of the OLE Period (up to 39 months).
Groups:
- Placebo 6-Month DB: Matching placebo (normal saline [0.9% NaCl]) was administered SC, QM, for 6 months during the 6-Month DB Period.
- All Givosiran: All participants treated with any amount of givosiran.
Arm/Group | Placebo 6-Month DB | Givosiran 2.5 mg/kg 6-Month DB | Placebo/Givosiran | Givosiran/Givosiran | All Givosiran
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/46 | 1/48 | 1/94
Serious Adverse Events (participants affected / at risk) | 4/46 | 10/48 | 17/46 | 20/48 | 37/94
Other Adverse Events (participants affected / at risk) | 37/46 | 43/48 | 44/46 | 47/48 | 91/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 6-Month DB (N=46) | Givosiran 2.5 mg/kg 6-Month DB (N=48) | Placebo/Givosiran (N=46) | Givosiran/Givosiran (N=48) | All Givosiran (N=94)
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pain management (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Administration site extravasation (General disorders) | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Catheter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Post procedural fever 1 (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Blood homocysteine increased (Investigations) | 0 | 0 | 2 | 0 | 2
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Device breakage (Product Issues) | 0 | 0 | 1 | 1 | 2
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 4
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Intrathecal pump insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Pain management (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Subclavian vein occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 6-Month DB (N=46) | Givosiran 2.5 mg/kg 6-Month DB (N=48) | Placebo/Givosiran (N=46) | Givosiran/Givosiran (N=48) | All Givosiran (N=94)
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 13 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 4 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 5 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 8 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 3 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 3 | 0 | 0 | 0
Lipase increased (Investigations) | 3 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 6 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 3 | 1 | 4
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 8 | 6 | 14
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 4 | 4 | 8
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 7 | 8 | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4 | 3 | 7
Nausea (Gastrointestinal disorders) | 0 | 0 | 12 | 22 | 34
Vomiting (Gastrointestinal disorders) | 0 | 0 | 8 | 7 | 15
Asthenia (General disorders) | 0 | 0 | 4 | 5 | 9
Fatigue (General disorders) | 0 | 0 | 13 | 12 | 25
Influenza like illness (General disorders) | 0 | 0 | 1 | 5 | 6
Injection site pain (General disorders) | 0 | 0 | 0 | 3 | 3
Oedema peripheral (General disorders) | 0 | 0 | 3 | 2 | 5
Pain (General disorders) | 0 | 0 | 4 | 3 | 7
Pyrexia (General disorders) | 0 | 0 | 6 | 6 | 12
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 3 | 1 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 4 | 2 | 6
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 3 | 5
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 3 | 3
Cystitis (Infections and infestations) | 0 | 0 | 3 | 3 | 6
Gastroenteritis (Infections and infestations) | 0 | 0 | 5 | 3 | 8
Influenza (Infections and infestations) | 0 | 0 | 5 | 4 | 9
Nasopharyngitis (Infections and infestations) | 0 | 0 | 11 | 14 | 25
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 3 | 6
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 12 | 7 | 19
Urinary tract infection (Infections and infestations) | 0 | 0 | 10 | 9 | 19
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 2 | 7
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 3 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4 | 4 | 8
Amylase increased (Investigations) | 0 | 0 | 3 | 4 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 4 | 7
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 5 | 7
Blood homocysteine increased (Investigations) | 0 | 0 | 1 | 3 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 3 | 5
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 2 | 5 | 7
Lipase increased (Investigations) | 0 | 0 | 6 | 7 | 13
Weight increased (Investigations) | 0 | 0 | 1 | 3 | 4
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 3 | 9
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 7 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 3 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 5 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 3 | 4
Headache (Nervous system disorders) | 0 | 0 | 7 | 13 | 20
Migraine (Nervous system disorders) | 0 | 0 | 1 | 6 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 3 | 1 | 4
Tremor (Nervous system disorders) | 0 | 0 | 2 | 3 | 5
Device occlusion (Product Issues) | 0 | 0 | 1 | 5 | 6
Depression (Psychiatric disorders) | 0 | 0 | 4 | 3 | 7
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 3 | 8
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 5
Hypertension (Vascular disorders) | 0 | 0 | 4 | 3 | 7
Injection site reaction (General disorders) | 0 | 0 | 14 | 16 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT03338816/Prot_002.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT03338816/SAP_003.pdf